CLINICAL TRIAL: NCT05844540
Title: L- Shape Symphyseal Autogenous Bone Block for Alveolar Ridge Augmentation in Anterior Maxilla and Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A015010222
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Atrophic Anterior Alveolar Ridge
Keywords: L- Shape autogenous bone block; symphysis; alveolar ridge augmentation; anterior maxilla and mandible

STUDY DESIGN:
Intervention Model Description: eleven partially edentulous patients seeking horizontal and vertical alveolar bone augmentation in the anterior maxilla or mandible were included in this study. For each patient, autogenous bone block was harvested from the symphysis, trimmed to L-shape and used to augment the anterior maxilla or mandible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- harvesting and augmentation of bone block (Other): autogenous bone block was harvested from the symphysis, trimmed to L-shape and used to augment the anterior maxilla or mandible horizontally and vertically.
  Interventions: Procedure: harvesting bone block; Procedure: Recipient site preparation; Procedure: implant insertion

INTERVENTIONS:
Procedure: harvesting bone block — Under local anesthesia, a sulcular incision was performed between lower right and left second premolars with an oblique incision distal to each one. After that, a full thickness mucoperiosteal flap was elevated to expose the anterior mandible including the entire symphysis and both mental nerves. By using piezo-surgery unit (Surgic Touch, Woodpecker, China), a rectangular bone block was harvested from the symphysis about 8mm in depth and 2mm wider than the recipient site to allow for contouring. The bone cuts were performed 5mm far from the apices of the anterior teeth, mental foramina, and inferior border of the mandible. Finally, thin curved osteotomes was used to detach the bone blocks. The harvested bone block was trimmed to form L-shape block and kept in normal saline. After hemostasis, the flap was closed with 4/0 vicryl interrupted sutures.
  Other Names: piezo-surgery block harvesting
Procedure: Recipient site preparation — At the maxillary recipient site, after induction of local anesthesia, a mid-crestal incision that continued in the sulcus for two teeth on either side of the defect with bilateral oblique incisions were performed. After that, the full thickness mucoperiosteal flap was elevated. While for mandibular recipient site, it was the same flap used for harvesting symphyseal bone block. For both upper or lower recipient sites, perforations (bone marrow penetration) were done to the recipient site by using a fissure surgical bur. The L-shape block graft was trimmed to obtain optimal adaptation to the recipient site, then it was fixed to the residual ridge with two 1.5mm self-tapping titanium screws. After attaining graft stability, any sharp edges were smoothed and any gap between the graft and underlying alveolar bone was filled with particulate bone curetted from the donner site.
Procedure: implant insertion — Implant insertion:
  After 6months, the surgical site was opened to remove fixation screws and insert dental implants, and the final restoration was done 4months after implant insertion.

SUMMARY:
the aim of this study was to assess both horizontal and vertical alveolar bone augmentation for sever atrophied anterior maxilla and mandible, using L- shape autogenous bone block harvested from the symphysis. eleven partially edentulous patients seeking horizontal and vertical alveolar bone augmentation in the anterior maxilla or mandible were included in this study. For each patient, autogenous bone block was harvested from the symphysis, trimmed to L-shape and used to augment the anterior maxilla or mandible horizontally and vertically. Horizontal and vertical bone gain was measured by CBCT immediate postoperative and at 6months after grafting.

DETAILED DESCRIPTION:
A total of 11 partially edentulous patients needing extensive horizontal and vertical bone augmentation in the anterior maxilla or mandible were included in this study. The patients were recruited from the Outpatient Clinic of Oral and Maxillofacial Department, Faculty of Dentistry, Mansoura University.

Before the surgical operation, all patients were informed about the treatment options, the nature of the operation, and the probable postoperative sequelae. An informed consent was signed from each patient.

Preoperative assessment

* Patients' medical status were carefully evaluated.
* A thorough intraoral examination was done to evaluate oral hygiene, occlusion, and mucosa that covers the recipient and donor sites.
* Preoperative CBCT was done for each patient to evaluate bone width and height in both the recipient and donor sites.

Surgical procedures Prophylactic antibiotic 600 mg Clindamycin (Clindam, Sigma, Egypt) was administered 1 hour before surgery. A thorough mouth rinsing using Chlorhexidine mouth wash (Hexitol, Adco, Egypt) for about 1 min was done immediately before surgery.

Harvesting procedure of the symphysis bone block:

Under local anesthesia, a sulcular incision was performed between lower right and left second premolars with an oblique incision distal to each one. After that, a full thickness mucoperiosteal flap was elevated to expose the anterior mandible including the entire symphysis and both mental nerves. By using piezo-surgery unit, a rectangular bone block was harvested from the symphysis about 8mm in depth and 2mm wider than the recipient site to allow for contouring. The bone cuts were performed 5mm far from the apices of the anterior teeth, mental foramina, and inferior border of the mandible. Finally, thin curved osteotomes was used to detach the bone blocks. The harvested bone block was trimmed to form L-shape block and kept in normal saline. After hemostasis, the flap was closed with 4/0 vicryl interrupted sutures.

Recipient site preparation:

At the maxillary recipient site, after induction of local anesthesia, a mid-crestal incision that continued in the sulcus for two teeth on either side of the defect with bilateral oblique incisions were performed. After that, the full thickness mucoperiosteal flap was elevated. While for mandibular recipient site, it was the same flap used for harvesting symphyseal bone block. For both upper or lower recipient sites, perforations (bone marrow penetration) were done to the recipient site by using a fissure surgical bur. The L-shape block graft was trimmed to obtain optimal adaptation to the recipient site, then it was fixed to the residual ridge with two 1.5mm self-tapping titanium screws. After attaining graft stability, any sharp edges were smoothed and any gap between the graft and underlying alveolar bone was filled with particulate bone curetted from the donner site. Finally, the flap was relaxed by periosteal incisions and blunt muscle dissection from the anterior maxilla or mandible to obtain a primary tension free closure using 4/0 vicryl interrupted and horizontal mattress sutures.

Postsurgical instructions:

Patients were instructed to avoid any wound trauma, and apply ice packs on the host and recipient surgical sites 20min/ hour for the first day after surgery. Proper oral hygiene should be maintained by mouth rinsing with chlorhexidine mouth wash 3times/ day for 1 week. Diclofenac potassium 50mg (Cataflam, Novartis, Switzerland) anti-inflammatory analgesic was prescribed as needed. Clindamycin 300mg twice daily was prescribed for 7days.

Implant insertion:

After 6months, the surgical site was opened to remove fixation screws and insert dental implants, and the final restoration was done 4months after implant insertion.

Evaluation: the patients were scheduled at 3days, 14days, 3months, and 6months postoperatively to evaluate:

ELIGIBILITY:
Inclusion Criteria:

* Missed one or more upper or lower anterior teeth.
* alveolar ridge with horizontal and vertical bone loss (class III according to Seibert et al(1983) classification).
* age 18 to 45 years.
* healthy oral mucosa, at least 3 mm keratinized mucosa.
* no systemic diseases or drugs that affect bone healing.
* no systemic or local conditions that contraindicate bone grafting or surgery.

Exclusion Criteria:

* Patients with disturbed occlusion, inadequate inter-arch space.
* patients with parafunction habits as bruxism or clenching.
* pregnancy.
* smokers.
* poor oral hygiene.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
numerical rating scale for pain measurement | 3 days post-surgery
  Pain intensity was measured at three days after surgery on a 0 to 10 numerical rating scale in which 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, and 10 = the worst pain imaginable.
infection and dehiscence of soft tissue | with in 6 months
  This was determined clinically by presence=1 or absence=0, of pus formation or graftb exposure.
questionnaire for sensory disturbance | with in 6 months
  This was assessed by patients' complaint (patient questionnaire) to determine any change in subjective sensation in the lower lip, chin and mental area. if there is pain or not. if there is numbness or not.
width of the alveolar ridge | immediate post-operative and after 6 months
  CBCT cross section view was used for evaluation of alveolar ridge width and preoperatively, immediate postoperative (within one week after grafting), and at 6 months after grafting.
height of the alveolar ridge | immediate post-operative and after 6 months
  CBCT cross section view was used for evaluation of alveolar height preoperatively, immediate postoperative (within one week after grafting), and at 6 months after grafting.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Eldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No